CLINICAL TRIAL: NCT04518761
Title: Predictive Modelling of the Intraoperative Train-of-Four (TOF) Ratio
Status: Recruiting | Type: Observational
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Other Study IDs: TOFPROS02
Record Dates: First submitted 2020-08-14; First posted 2020-08-19 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Analyse Neuromuscular Monitoring for Developing a Model to Predict TOF Ratio During Anesthesia
MeSH Terms: interventions — Elective Surgical Procedures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prospective group
  Interventions: Procedure: Elective surgery
- Retrospective group
  Interventions: Procedure: Elective surgery

INTERVENTIONS:
Procedure: Elective surgery — Any patient who needs to undergo an elective surgery.

SUMMARY:
Neuromuscular Blocking Agents (NMBAs) are routinely administered to patients in a multiplicity o anaesthetic settings in order to paralyze and impede (re)active muscular contraction. The availability of monitoring devices allowing an accurate measurement fo the degree of neuromuscular block during anesthesia has raised the standards for a proper evidence-based use of NMBAs.

For this purpose, one of the most widely used methods is the Train of Four (TOF): transcutaneous application of a series of 4 square-wave supra-maximal electrical stimuli over the course of a nerve of choice (most commonly the ulnar nerve). These are applied at a frequency of 2Hz, and each with a duration of 0.2ms. These stimuli elicit a motor response on the adductor pollicis muscle, which on its turn dictates the adduction of the thumb. The acceleration of this movement can be followed by means of an uni/multi-directional accelerometer attached to the thumb. The ratio of the acceleration of the 4th and 1st elicited contractions is called the TOF-Ratio - a clinically and scientifically established method of assessing neuromuscular block recovery. A value of 1 translates a full recovery of the muscular function of a patient. In modern Anesthesia, the bar for deeming a recovery as adequate has been set at a minimum of a TOF-ratio of >0.9, with some authors advocating a ratio of 1 as the only acceptable and complications avoiding result.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 years old and above) receiving General Anesthesia for noncardiac surgery requiring the use of a neuromuscular blocking agent.
* Administration of General Anesthesia by means of Total Intravenous Anesthesia technique.
* Use of Rocuronium as a neuromuscular blocking agent.

Exclusion Criteria:

* Use of different types of neuromuscular blocking agents for the same patient within the same surgical procedure
* Known Neuromuscular diseases/syndromes judged to condition accurate neuromuscular monitoring.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (18 years old and above) receiving General Anesthesia for noncardiac surgery requiring the use of a neuromuscular blocking agent.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
TOF-ratio | 1 day
  Train of four percentage

SECONDARY OUTCOMES:
TOF-count | 1 day
  Train of four count

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - UZ Brussel, Jette, Brussels Capital
  - AZ Sint Jan, Bruges, WV

IPD SHARING:
Plan to Share IPD: Undecided
Publication via medical article.

REFERENCES:
- [Derived] Verdonck M, Carvalho H, Fuchs-Buder T, Brull SJ, Poelaert J. Machine learning based analysis and detection of trend outliers for electromyographic neuromuscular monitoring. J Clin Monit Comput. 2024 Oct;38(5):1163-1173. doi: 10.1007/s10877-024-01141-6. Epub 2024 Apr 4. PMID 38573367
- [Derived] Carvalho H, Verdonck M, Eleveld DJ, Ramirez D, D'Haese J, Flamee P, Geerts L, Wylleman J, Cools W, Barbe K, Struys MMRF, Poelaert J. Neuromuscular end-point predictive capability of published rocuronium pharmacokinetic/pharmacodynamic models: An observational trial. J Clin Anesth. 2023 Nov;90:111225. doi: 10.1016/j.jclinane.2023.111225. Epub 2023 Aug 3. PMID 37542918